CLINICAL TRIAL: NCT03509038
Title: Urodynamic Evaluation of Incontinent Obese Women Before and After Weight Reduction by Bariatric Surgery : What Urodynamic Healing Factors? BUDI (Bariatric UroDynamic Improvement)
Brief Title: BUDI (Bariatric UroDynamic Improvement)
Acronym: BUDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02121-52
Record Dates: First submitted 2018-03-14; First posted 2018-04-26 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Urinary Incontinence; Obesity; Urodynamics; Quality of Life
MeSH Terms: conditions — Urinary Incontinence; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urinary incontinence before bariatric surgery (Experimental): All patients with urinary incontinence before bariatric surgery will be addressed for a urodynamic exam
  Interventions: Other: Exploratory pathophysiology Study

INTERVENTIONS:
Other: Exploratory pathophysiology Study — Urodynamic tests before and after bariatric surgery in obese incontinent women before and after bariatric surgery

SUMMARY:
In the population of obese women, the prevalence of urinary incontinence (UI) is around 70%. It was shown in the literature that weight loss by bariatric surgery allowed a significant improvement in the symptoms and impact on the quality of life of the IU. However, no prognostic factor for recovery has yet been identified and the pathophysiological mechanisms underpinning this improvement are not fully elucidated.

The main objective of this study is to highlight the urodynamic changes associated with the improvement of the symptom and quality of life scores in a population of incontinent obese women before and after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

The research protocol will be proposed to all patients requiring bariatric surgery (gastric bypass or sleeve gastrectomy) and describing urinary incontinence according to the definition of the International Continence Society (ICS)

Exclusion Criteria:

* minors under the age of 18
* pregnant or lactating women
* women not speaking French (important to understand and respond to questionnaires)
* women who have not given their written consent
* neurological diseases,
* patients who have benefited from urinary incontinence surgery, prolapse treatment or pelvic surgery at risk of urodynamic modifications (extensive resection of deep endometriosis, pelvic wound surgery, pelvic radiation therapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Urodynamic changes after bariatric surgery in obese incontinent women | 24 months
  to highlight the changes in urodynamic vesical pressure (cmH2O) associated with the improvement of urinary incontinence after bariatric surgery
Urodynamic changes after bariatric surgery in obese incontinent women | 24 months
  to highlight the changes in urodynamic vesical sensations (cmH2O) associated with the improvement of urinary incontinence after bariatric surgery
Urodynamic changes after bariatric surgery in obese incontinent women | 24 months
  to highlight the changes in urodynamic bladder-to-urethra pressure transmission (%) with cough associated with the improvement of urinary incontinence after bariatric surgery
Urodynamic changes after bariatric surgery in obese incontinent women | 24 months
  to highlight the changes in urodynamic maximum urethral cloture pressure (cmH2O) associated with the improvement of urinary incontinence after bariatric surgery

SECONDARY OUTCOMES:
Urinary incontinence symptom improvement after bariatric surgery | 24 months
  Changes in ICIQ-SF (International Consultation on Incontinence Questionnaire - Short Form) scores (assessing frequency and quantity of urinary loss, ranging from 0 to 21) after weight loss in incontinent obese women
Quality of life improvement after bariatric surgery | 24 months
  Measuring changes in Quality of life after weight loss with the Contilife questionnaire which specifically measures the impact of urinary incontinence on quality of life : activity of daily life
Quality of life improvement after bariatric surgery | 24 months
  Measuring changes in Quality of life after weight loss with the Contilife questionnaire which specifically measures the impact of urinary incontinence on quality of life : self-image and emotional impact and sexuality)
Quality of life improvement after bariatric surgery | 24 months
  Measuring changes in Quality of life after weight loss with the Contilife questionnaire which specifically measures the impact of urinary incontinence on quality of life : sexuality

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Cécile Pizzoferrato, MD, PhD, Principal Investigator — University hospital of Caen
Locations (1):
- Pizzoferato, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided
study protocol statistical analysis plan informed consent form analytic code clinical study report

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Legendre G, Fritel X, Capmas P, Pourcelot AG, Fernandez H. [Urinary incontinence and obesity]. J Gynecol Obstet Biol Reprod (Paris). 2012 Jun;41(4):318-23. doi: 10.1016/j.jgyn.2012.02.007. Epub 2012 Apr 17. French. PMID 22516035
- [Background] Sandvik H, Hunskaar S, Seim A, Hermstad R, Vanvik A, Bratt H. Validation of a severity index in female urinary incontinence and its implementation in an epidemiological survey. J Epidemiol Community Health. 1993 Dec;47(6):497-9. doi: 10.1136/jech.47.6.497. PMID 8120507
- [Background] Subak LL, Richter HE, Hunskaar S. Obesity and urinary incontinence: epidemiology and clinical research update. J Urol. 2009 Dec;182(6 Suppl):S2-7. doi: 10.1016/j.juro.2009.08.071. PMID 19846133
- [Background] Elia G, Dye TD, Scariati PD. Body mass index and urinary symptoms in women. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(6):366-9. doi: 10.1007/pl00004043. PMID 11795637
- [Background] Luber KM. The definition, prevalence, and risk factors for stress urinary incontinence. Rev Urol. 2004;6 Suppl 3(Suppl 3):S3-9. PMID 16985863
- [Background] Neels JG, Olefsky JM. Inflamed fat: what starts the fire? J Clin Invest. 2006 Jan;116(1):33-5. doi: 10.1172/JCI27280. PMID 16395402
- [Background] Agur W, Rizk DE. Obesity and urinary incontinence in women: is the black box becoming grayer? Int Urogynecol J. 2011 Mar;22(3):257-8. doi: 10.1007/s00192-010-1293-z. Epub 2010 Oct 6. No abstract available. PMID 20924556
- [Background] Lose G, Tanko A, Colstrup H, Andersen JT. Urethral sphincter electromyography with vaginal surface electrodes: a comparison with sphincter electromyography recorded via periurethral coaxial, anal sphincter needle and perianal surface electrodes. J Urol. 1985 May;133(5):815-8. doi: 10.1016/s0022-5347(17)49238-x. PMID 4039373
- [Background] Sapsford RR, Hodges PW. Contraction of the pelvic floor muscles during abdominal maneuvers. Arch Phys Med Rehabil. 2001 Aug;82(8):1081-8. doi: 10.1053/apmr.2001.24297. PMID 11494188
- [Background] Banerjea R, Findley PA, Sambamoorthi U. Disparities in preventive care by body mass index categories among women. Women Health. 2008;47(4):1-17. doi: 10.1080/03630240802099261. PMID 18843937
- [Background] Elliott V, de Bruin ED, Dumoulin C. Virtual reality rehabilitation as a treatment approach for older women with mixed urinary incontinence: a feasibility study. Neurourol Urodyn. 2015 Mar;34(3):236-43. doi: 10.1002/nau.22553. Epub 2014 Jan 10. PMID 24415577
- [Result] Chen CC, Gatmaitan P, Koepp S, Barber MD, Chand B, Schauer PR, Brethauer SA. Obesity is associated with increased prevalence and severity of pelvic floor disorders in women considering bariatric surgery. Surg Obes Relat Dis. 2009 Jul-Aug;5(4):411-5. doi: 10.1016/j.soard.2008.10.006. Epub 2008 Oct 29. PMID 19136310
- [Result] Knepfler T, Valero E, Triki E, Chilintseva N, Koensgen S, Rohr S. Bariatric surgery improves female pelvic floor disorders. J Visc Surg. 2016 Apr;153(2):95-9. doi: 10.1016/j.jviscsurg.2015.11.011. Epub 2015 Dec 8. PMID 26678846
- [Result] Kuruba R, Almahmeed T, Martinez F, Torrella TA, Haines K, Nelson LG, Gallagher SF, Murr MM. Bariatric surgery improves urinary incontinence in morbidly obese individuals. Surg Obes Relat Dis. 2007 Nov-Dec;3(6):586-90; discussion 590-1. doi: 10.1016/j.soard.2007.08.007. Epub 2007 Oct 18. PMID 17950043
- [Result] Burgio KL, Richter HE, Clements RH, Redden DT, Goode PS. Changes in urinary and fecal incontinence symptoms with weight loss surgery in morbidly obese women. Obstet Gynecol. 2007 Nov;110(5):1034-40. doi: 10.1097/01.AOG.0000285483.22898.9c. PMID 17978117
- [Result] Richter HE, Kenton K, Huang L, Nygaard I, Kraus S, Whitcomb E, Chai TC, Lemack G, Sirls L, Dandreo KJ, Stoddard A. The impact of obesity on urinary incontinence symptoms, severity, urodynamic characteristics and quality of life. J Urol. 2010 Feb;183(2):622-8. doi: 10.1016/j.juro.2009.09.083. Epub 2009 Dec 16. PMID 20018326
- [Result] Richter HE, Creasman JM, Myers DL, Wheeler TL, Burgio KL, Subak LL; Program to Reduce Incontinence by Diet and Exercise (PRIDE) Research Group. Urodynamic characterization of obese women with urinary incontinence undergoing a weight loss program: the Program to Reduce Incontinence by Diet and Exercise (PRIDE) trial. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Dec;19(12):1653-8. doi: 10.1007/s00192-008-0694-8. Epub 2008 Aug 5. PMID 18679560
- [Result] Nathan PA, Keniston RC, Myers LD, Meadows KD. Obesity as a risk factor for slowing of sensory conduction of the median nerve in industry. A cross-sectional and longitudinal study involving 429 workers. J Occup Med. 1992 Apr;34(4):379-83. PMID 1564575
- [Result] Bump RC, Sugerman HJ, Fantl JA, McClish DK. Obesity and lower urinary tract function in women: effect of surgically induced weight loss. Am J Obstet Gynecol. 1992 Aug;167(2):392-7; discussion 397-9. doi: 10.1016/s0002-9378(11)91418-5. PMID 1497041
- [Result] Romero-Talamas H, Unger CA, Aminian A, Schauer PR, Barber M, Brethauer S. Comprehensive evaluation of the effect of bariatric surgery on pelvic floor disorders. Surg Obes Relat Dis. 2016 Jan;12(1):138-43. doi: 10.1016/j.soard.2015.08.499. Epub 2015 Aug 13. PMID 26686304
- [Result] Amarenco G, Ismael SS, Lagauche D, Raibaut P, Rene-Corail P, Wolff N, Thoumie P, Haab F. Cough anal reflex: strict relationship between intravesical pressure and pelvic floor muscle electromyographic activity during cough. Urodynamic and electrophysiological study. J Urol. 2005 Jan;173(1):149-52. doi: 10.1097/01.ju.0000147305.00443.df. PMID 15592060
- [Result] Townsend MK, Curhan GC, Resnick NM, Grodstein F. BMI, waist circumference, and incident urinary incontinence in older women. Obesity (Silver Spring). 2008 Apr;16(4):881-6. doi: 10.1038/oby.2008.14. Epub 2008 Feb 14. PMID 18379564
- [Result] Deffieux X, Hubeaux K, Porcher R, Ismael SS, Raibaut P, Amarenco G. Pelvic floor muscle activity during coughing: altered pattern in women with stress urinary incontinence. Urology. 2007 Sep;70(3):443-7; discussion 447-8. doi: 10.1016/j.urology.2007.03.084. PMID 17905093